CLINICAL TRIAL: NCT06179940
Title: Evaluation of the Effect of Food Selectivity Intervention in Children With Autism Spectrum Disorders.
Brief Title: Food Selectivity Protocol for Children With Autism Spectrum Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Messina, Italy (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2023-009
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; children; food selectivity
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food selectivity group (1) in pairs (Experimental): 15 Children in the experimental group who will undergo the treatment perform the procedure in pairs.
  Interventions: Other: Pairwise food selectivity protocol
- Food selectivity Group (2) in individual mode (Experimental): 15 Children in the comparator group who will undergo the treatment perform the procedure in individual mode.
  Interventions: Other: Individual food selectivity protocol

INTERVENTIONS:
Other: Pairwise food selectivity protocol — Overall, the intervention aims to gradually expose the child to various foods, starting with familiarization, progressing to exposure without pressure, and finally, shaping positive behaviors using reinforcement and observing reactions to different food items. The experimental group will conduct the protocol activity in pairs.
  Arms: Food selectivity group (1) in pairs
Other: Individual food selectivity protocol — Overall, the intervention aims to gradually expose the child to various foods, starting with familiarization, progressing to exposure without pressure, and finally, shaping positive behaviors using reinforcement and observing reactions to different food items. The control group will conduct the activity individually.
  Arms: Food selectivity Group (2) in individual mode

SUMMARY:
Food selectivity is a common challenge among children with Autism Spectrum Disorder (ASD), with significant impacts on their nutrition and well-being. The main purpose of this study is to promote children's active participation in mealtime routines and encourage experimentation with new foods through an approach that emphasizes joy and serenity during mealtimes. The study will involve children with ASD between the ages of 4 and 10 years, of both sexes. Food selectivity will be assessed through interviews with parents and the use of specially created cards.

The protocol will include 45-minute sessions, twice a week, for a total of 48 sessions. During these sessions, two plates, a list of foods previously agreed upon with the parents, and the foods needed for each session will be used. The sessions will take place in an environment called "Home Lab"a specially set up as if it were a kitchen to reproduce a home atmosphere.

DETAILED DESCRIPTION:
Food selectivity training is divided into three steps. Step 1- Pairing in the kitchen. Propose highly enjoyed activities to the child in the kitchen. Criterion for moving to step 2: Child stays in the kitchen to play for 5 minutes for 3 consecutive sessions.

Indicate the minutes of playing in the kitchen.

Step 2 Food selectivity training is divided into three steps. Step 1- Pairing in the kitchen. Propose highly enjoyed activities to the child in the kitchen. Criterion for moving to step 2: Child stays in the kitchen to play for 5 minutes for 3 consecutive sessions.

Indicate the minutes of playing in the kitchen. Step 2 At the beginning of the session prepare two identical plates, in each plate there will be 6 foods, arranged in the same way. Place them on the table in the kitchen.

Training

* Transition living room (carpet) - kitchen (table)
* The child is participating in a welcome game with the operator;
* the operator waits 30 sec for the child to spontaneously interact with him: he approaches, stands up and tries to take the operator's hand
* Immediately afterwards, the operator accompanies the child to the kitchen.
* If the child does NOT spontaneously interact with the operator within 30 sec then says, "Let's go."
* If the child does NOT follow the operator's prompt within 30 sec, the operator repeats the prompt once. If the child does not follow the prompt the session will be postponed until the next day.
* NB: If the latter situation occurs (the child does not follow the prompt and therefore the session is postponed) note what happened.
* Procedure
* the operator sits next to the child(ren);
* the operator interacts with the food, without eating it (e.g., touches it, smells it ...).
* During the session, the operator maintains a positive expression, talks about general topics not related to food.
* the practitioner does NOT give any prompt to the child to taste or eat the food.
* The child can walk away at any time. Criterion for moving to stage 3: Child remains seated with plate in front of him/her for 30 sec without emitting problem behaviors for 3 consecutive sessions.

Indicate the time (seconds) in which the child remains sitting with the plate in front of him without stress.

Step 3 - Shaping

- At the beginning of the session prepare two identical plates, in each plate there will be 6 foods, arranged in the same way. Place them on the table in the kitchen.

* Operator inserts comments about the food (e.g., "these carrots are delicious").
* The operator prepares a small container with small pieces with the child's favorite food. The favorite food should only be available at the shaping stage. The container with the favorite food must be out of the child's reach but must be visible to him. The favorite food should not be in the saucer, even in stage 2.
* The caregiver observes any food-related behavior of the child (for example: looks at it, touches it ...). If the child emits any food-related behavior the operator immediately reinforces by praising it and giving it a piece of the favorite food.

The operator defines the target behaviors to be reinforced.

* If the child does not emit any target behavior for more than 15 sec, the operator selects a different target behavior.
* If the child shows any negative emotion at any time during the session, the operator immediately changes the target behavior. To encourage the emergence of different behaviors, the practitioner will differentially reinforce the child's responses. The experimental group will conduct the protocol activity in pairs, and the control group individually.

ELIGIBILITY:
Inclusion Criteria:

* Food selectivity upon parental referral
* diagnosis of autism

Exclusion Criteria:

* presence of other medical disorders

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-07-17 (Estimated)

PRIMARY OUTCOMES:
Brief Autism Mealtime Behavior Inventory (BAMBI) | The test need approximately 10 minutes
  the Bambi measures food selectivity, disruptive behavior, food refusal and rigidity at mealtime
  The 18-item Brief Autism Mealtime Behavior Inventory (BAMBI) is a parent-report questionnaire that was created to identify mealtime habits unique to kids with ASD.
  The BAMBI is rated on a Likert scale of 1 to 5, where 1 represents "never" occurring behavior during mealtime and 5 represents "always" occurring behavior. For four of the items that rate constructive mealtime behaviors, reversed scoring is applied. The sum of the 18 elements is used to create the total frequency score, with higher scores indicating more issues with behavior during meals.
inventory of food preferences | The test need approximately 20 minutes
  The food preference inventory includes a list of foods that is submitted to the parent. Asked how often the food is consumed by the child and family
general assessment checklist | The test need approximately 15 minutes
  the general assessment includes a personal data sheet, the section relating to nutrition and therefore to the dietary regime, the type of selectivity and dysfunctional behaviours. Finally there is the adaptive functioning card relating to autonomy during meals.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Istituto per la Ricerca e l'Innovazione Biomedica
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piazza CC, Patel MR, Santana CM, Goh HL, Delia MD, Lancaster BM. An evaluation of simultaneous and sequential presentation of preferred and nonpreferred food to treat food selectivity. J Appl Behav Anal. 2002 Fall;35(3):259-70. doi: 10.1901/jaba.2002.35-259. PMID 12365739
- [Background] Esposito M, Mirizzi P, Fadda R, Pirollo C, Ricciardi O, Mazza M, Valenti M. Food Selectivity in Children with Autism: Guidelines for Assessment and Clinical Interventions. Int J Environ Res Public Health. 2023 Mar 14;20(6):5092. doi: 10.3390/ijerph20065092. PMID 36982001
- [Background] Peterson KM, Piazza CC, Ibanez VF, Fisher WW. Randomized controlled trial of an applied behavior analytic intervention for food selectivity in children with autism spectrum disorder. J Appl Behav Anal. 2019 Oct;52(4):895-917. doi: 10.1002/jaba.650. PMID 31642526